CLINICAL TRIAL: NCT00419744
Title: A Phase IIIB, 12-Month, Double-blind, Double-dummy,Randomised, Parallel-group, Multicentre Exacerbation Study of SYMBICORT® pMDI 160/4.5 μg x 2 Actuations Twice-daily and 80/4.5 μg x 2 Actuations Twice-daily Compared to Formoterol Turbuhaler® 4.5 μg x 2 Inhalations Twice-daily in COPD Subjects
Brief Title: A Comparison of SYMBICORT® pMDI With Formoterol Turbuhaler® in Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D589CC00003
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol (SYMBICORT) pMDI
Drug: Formoterol Turbuhaler

SUMMARY:
The purpose of this study is to determine if SYMBICORT® delivered via a pressurized metered-dose inhaler, referred to as a pMDI, is effective in preventing COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* A current clinical diagnosis of COPD with COPD symptoms for more than 2 years
* Current smoker or smoking history of 10 or more pack years (1 pack year = 20 cigarettes smoked per day for one year)
* A history of at least 1 COPD exacerbations requiring a course of steroids and/or antibiotics within 1-12 months before the first visit

Exclusion Criteria:

* A history of asthma at or after 18 years of age
* A history of allergic rhinitis at or after 18 years of age
* Subjects taking oral steroids
* Any significant disease or disorder that may jeopardize a subject's safety

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultquist, MD, Study Director — AstraZeneca
Locations (140):
- United States (92):
  - Research Site, Jasper, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Foothill Ranch, California
  - Research Site, Fullerton, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Los Banos, California
  - Research Site, Mission Viejo, California
  - Research Site, Pismo Beach, California
  - Research Site, Rancho Cordova, California
  - Research Site, Rancho Mirage, California
  - Research Site, Riverside, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Sepulveda, California
  - Research Site, Torrance, California
  - Research Site, Englewood, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Stanford, Connecticut
  - Research Site, DeLand, Florida
  - Research Site, Opa-locka, Florida
  - Research Site, Orange City, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Saint Cloud, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Council Bluffs, Iowa
  - Research Site, Witchita, Kansas
  - Research Site, Marrero, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Waltham, Massachusetts
  - Research Site, Chesterfield, Missouri
  - Research Site, Florissant, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Springfield, New Jersey
  - Research Site, Bronxville, New York
  - Research Site, Elmira, New York
  - Research Site, Larchmont, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Chardon, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Beaver, Pennsylvania
  - Research Site, Bensalem, Pennsylvania
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Landsdale, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warminster, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Prosperity, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Fayetteville, Tennessee
  - Research Site, Boerne, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
- Argentina (10):
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Nueve de Julio, Buenos Aires
  - Research Site, Ramos Mejía, Buenos Aires
  - Research Site, Vicente López, Buenos Aires
  - Research Site, Corrientes, Corrientes Province
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, San Juan, San Juan Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
- Brazil (10):
  - Research Site, Fortaleza, Ceará
  - Research Site, Goiânia, Goiás
  - Research Site, Curitiba, Paraná
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porta Alegre, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Florian�polis, Santa Catarina
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Chile (3):
  - Research Site, Valparaíso, Región de Valparaíso
  - Research Site, Rancagua, Región del Libertador General Bernardo O’Higgins
  - Research Site, Santiago, RM
- Colombia (3):
  - Research Site, Medillin, Antioquia
  - Research Site, Barranquilla, Atl�ntico
  - Research Site, Bogota Dc, Cundianmarca
- Research Site, Guadalajara, Jalisco, Mexico
- Peru (4):
  - Research Site, Lima, Lima Province
  - Research Site, Jesus Maria, Lima region
  - Research Site, San Borja, Lima region
  - Research Site, Surco, Lima region
- South Africa (16):
  - Research Site, Belvilee, Cape Town
  - Research Site, Tygerberg, Cape Town
  - Research Site, Port Elizabeth, E Cape
  - Research Site, Korsten, Port Elizabeth
  - Research Site, Groenkloof, Pretoria
  - Research Site, Thaba Tswane, Pretoria
  - Research Site, Cape Town, South Africa
  - Research Site, Durban, South Africa
  - Research Site, Bloemfontein
  - Research Site, Boksburg
  - Research Site, Centurion
  - Research Site, eManzimtoti
  - Research Site, Humansdorp
  - Research Site, Pretoria
  - Research Site, Pretoria West
  - Research Site, Roodepoort
- Research Site, Distrito Capital, Miranda, Venezuela

REFERENCES:
- [Derived] Bafadhel M, Peterson S, De Blas MA, Calverley PM, Rennard SI, Richter K, Fageras M. Predictors of exacerbation risk and response to budesonide in patients with chronic obstructive pulmonary disease: a post-hoc analysis of three randomised trials. Lancet Respir Med. 2018 Feb;6(2):117-126. doi: 10.1016/S2213-2600(18)30006-7. Epub 2018 Jan 10. PMID 29331313
- [Derived] Jenkins CR, Postma DS, Anzueto AR, Make BJ, Peterson S, Eriksson G, Calverley PM. Reliever salbutamol use as a measure of exacerbation risk in chronic obstructive pulmonary disease. BMC Pulm Med. 2015 Aug 21;15:97. doi: 10.1186/s12890-015-0077-0. PMID 26293575
- [Derived] Make BJ, Eriksson G, Calverley PM, Jenkins CR, Postma DS, Peterson S, Ostlund O, Anzueto A. A score to predict short-term risk of COPD exacerbations (SCOPEX). Int J Chron Obstruct Pulmon Dis. 2015 Jan 27;10:201-9. doi: 10.2147/COPD.S69589. eCollection 2015. PMID 25670896
- [Derived] Sharafkhaneh A, Southard JG, Goldman M, Uryniak T, Martin UJ. Effect of budesonide/formoterol pMDI on COPD exacerbations: a double-blind, randomized study. Respir Med. 2012 Feb;106(2):257-68. doi: 10.1016/j.rmed.2011.07.020. Epub 2011 Oct 26. PMID 22033040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomized on 02 January 2007. The last patient completed study on 27 August 2009. The study randomized patients in the United States and Mexico (93 investigational sites), South America (48 investigational sites), and South Africa (20 investigational sites).
Pre-assignment Details: The study consisted of an initial screening visit (Visit 1) and 2-week run-in enrollment visits (Visits 2 and 3) prior to being randomized to 1 of 3 treatment groups
Groups:
- SYM 160/4.5 X 2 BID: SYMBICORT pMDI (budesonide/formoterol) 160/4.5 μg (delivered dose) per actuation, 2 actuations administered twice daily (BID)
- SYM 80/4.5 X 2 BID: SYMBICORT pMDI (budesonide/formoterol) 80/4.5 μg (delivered dose) per actuation, 2 actuations administered BID
- FOR 4.5 X 2 BID: Formoterol Turbuhaler 4.5 μg x 2 inhalations BID
Period: Overall Study
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Started | 407 | 408 | 404
Completed | 290 | 290 | 271
Not Completed | 117 | 118 | 133
Not completed — Adverse Event | 39 | 40 | 50
Not completed — Withdrawal by Subject | 45 | 49 | 52
Not completed — Lost to Follow-up | 8 | 10 | 6
Not completed — Protocol Violation | 4 | 7 | 8
Not completed — Randomized in error | 9 | 6 | 7
Not completed — Moving out of state | 2 | 0 | 1
Not completed — Physician Decision | 10 | 5 | 6
Not completed — Spirometry mouthpiece issues | 0 | 1 | 2
Not completed — Incorrect medication kit dispensed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID | Total
Number analyzed (Participants) | 407 | 408 | 403 | 1218
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (9.4) | 62.8 (9.22) | 62.5 (9.36) | 63.0 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 144 | 174 | 463
  Male | 262 | 264 | 229 | 755

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Per Patient-treatment Year
Description: Number of COPD-related exacerbations per patient-treatment year. COPD-related exacerbation was defined as worsening COPD that required a course of oral steriods for treatment and/or hospitalization.
Time Frame: 12 months
Measure: Number; unit: Exacerbations
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 404 | 403 | 403
Exacerbations | 0.75 | 0.84 | 1.14

2. Secondary Outcome: Pre-dose Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in pre-dose FEV1 from baseline to the average of the randomized treatment period, as calculated by averaging treatment period FEV1 values and subtracting the pre-dose value.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 399 | 399 | 399
Liters (L) | 0.07 (0.18) | 0.07 (0.17) | 0.04 (0.17)

3. Secondary Outcome: Morning Peak Expiratory Flow (PEF)
Description: Change in morning PEF from baseline to the average of the randomized treatment period, as calculated by averaging treatment period PEF values and subtracting the baseline morning PEF value.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 399 | 397 | 389
L/min | 19.82 (37.96) | 19.61 (38.83) | 15.81 (41.43)

4. Secondary Outcome: Evening PEF
Description: Change in evening PEF from baseline to the average of the randomized treatment period, as calculated by averaging treatment period PEF values and subtracting the baseline evening PEF value.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 400 | 397 | 393
L/min | 17.62 (37.86) | 17.77 (37.67) | 14.08 (41.13)

5. Secondary Outcome: Dyspnea Symptom Scores
Description: Change from baseline of Dyspnea symptoms evaluated using the breathlessness diary, a 5-point Likert-type scale, ranging from 0 to 4 with higher scores indicating a more severe manifestation of the Dyspnea symptom. Change from baseline was calculated by averaging treatment period Dyspnea scores and subtracting the baseline Dyspnea scores.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 401 | 400 | 398
Scores on a scale | -0.30 (0.65) | -0.29 (0.70) | -0.24 (0.67)

6. Secondary Outcome: Use of Rescue Medication
Description: Change from baseline in the use of beta-2 agonists, as calculated by averaging treatment period inhalations per day and subtracting the baseline number of inhalations per day.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of inhalations
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 401 | 401 | 399
Number of inhalations | -1.21 (3.57) | -1.03 (3.74) | -0.28 (3.60)

7. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Score
Description: Change from baseline in the SGRQ overall score, as calculated by averaging treatment period SGRQ scores and subtracting the baseline SGRQ scores. The SGRQ contains 3 domains: Symptoms (distress due to respiratory symptoms, 8 questions), Activity (disturbance of physical activity, 16 questions), and Impacts (overall impact on daily life and well-being, 26 questions). Lower scores are associated with less severe symptoms.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 375 | 366 | 357
Scores on a scale | -6.23 (14.72) | -5.00 (16.10) | -5.71 (15.31)

8. Primary Outcome: Rate of Exacerbations Per Subject-year
Description: Rate of exacerbations per subject-year
Time Frame: 12 months
Measure: Number; unit: Rate
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Number analyzed (Participants) | 404 | 403 | 403
Rate | 0.639 | 0.745 | 1.029

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SYM 160/4.5 X 2 BID | SYM 80/4.5 X 2 BID | FOR 4.5 X 2 BID
Serious Adverse Events (participants affected / at risk) | 79/407 | 61/408 | 73/403
Other Adverse Events (participants affected / at risk) | 193/407 | 177/408 | 176/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYM 160/4.5 X 2 BID (N=407) | SYM 80/4.5 X 2 BID (N=408) | FOR 4.5 X 2 BID (N=403)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 6 | 3 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 3
Cardiac Failure Congestive (Cardiac disorders) | 3 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 2
Cor Pulmonale (Cardiac disorders) | 0 | 1 | 2
Cardiac Failure Acute (Cardiac disorders) | 2 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 2 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial Tachycardia (Cardiac disorders) | 0 | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 13 | 4 | 7
Bronchitis (Infections and infestations) | 0 | 0 | 3
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bronchitis Bacterial (Infections and infestations) | 1 | 0 | 1
Dengue Fever (Infections and infestations) | 0 | 0 | 1
Enterocolitis Bacterial (Infections and infestations) | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia Viral (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Drug Toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Collapse Of Lung (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation Of Joint Prosthesis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Small Cell Lung Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Anxiety Disorder (Psychiatric disorders) | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Renal Aneurysm (Renal and urinary disorders) | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal Mass (Renal and urinary disorders) | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 32 | 33 | 34
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Accelerated Hypertension (Vascular disorders) | 0 | 0 | 1
Arterial Thrombosis Limb (Vascular disorders) | 0 | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1
Iliac Artery Occlusion (Vascular disorders) | 0 | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Intermittent Claudication (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SYM 160/4.5 X 2 BID (N=407) | SYM 80/4.5 X 2 BID (N=408) | FOR 4.5 X 2 BID (N=403)
Nasopharyngitis (Infections and infestations) | 31 | 35 | 41
Bronchitis (Infections and infestations) | 37 | 32 | 25
Influenza (Infections and infestations) | 29 | 26 | 25
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 18 | 23 | 17
Viral Upper Respiratory Tract Infection (Infections and infestations) | 21 | 13 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 21 | 18 | 21
Headache (Nervous system disorders) | 56 | 46 | 43
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 57 | 46 | 68
Hypertension (Vascular disorders) | 21 | 16 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may use the Multi-Center Study Results and the Site Data for the limited purpose of his or her own research and academic analysis until the earlier of the publication of the first Multi-center Publication and the second anniversary of the completion of the Multi-center Study at all participating sites.